CLINICAL TRIAL: NCT01875497
Title: Effect of Vitis Vinifera Extract on Oxidative Stress, Inflammatory Biomarkers and Hormones in High Trained Subjects After Resting and Intensive Physical Activity.
Brief Title: Effect of Vitis Vinifera Extract on Oxidative Stress, Inflamatory Biomarkers and Hormones in High Trained Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Josely Correa Koury, PhD, Rio de Janeiro State University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: E26-103.011/2012
Record Dates: First submitted 2013-06-05; First posted 2013-06-11 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Athletic Injuries
Keywords: athletes, polyphenols, nutrition, oxidative stress
MeSH Terms: conditions — Athletic Injuries | interventions — whole grape extract; Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dietary Supplement (Experimental): Before the exercise, the individuals intake only one capsule with 205 mg of the grape fruit extract in capsule with 205 mg.
  Interventions: Dietary Supplement: grape fruit (vitis vinifera) extract in capsule with 205 mg

INTERVENTIONS:
Dietary Supplement: grape fruit (vitis vinifera) extract in capsule with 205 mg — Before the exercise the indivuduals intake only one capsule of the grape fruit extract with 205 mg. This dosage is free of contraindications according to others studies.

SUMMARY:
There is evidence that intense physical activity has a potential effect on thrombotic events due to catecholamine release. The hormones leptin and adiponectin have been used as markers of cardiovascular risk, but they are few and contradictory studies that relate physical training intensity and duration of high plasma concentrations of these hormones. The use of antioxidants, such as proanthocyanidins present in grapes, may help in reducing the undesirable effects of intense training.

DETAILED DESCRIPTION:
Fifty four Brazilian healthy military without hyperglycemia, diabetes mellitus and endocrine disease were enrolled in this study. All subjects were high physically military trained. The Ethical Committee of the Universidade do Estado do Rio de Janeiro in Brazil (COEP008/2011) approved the study protocol. Informed consent was obtained from each subject after explanation of purpose and risks of all procedures used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy physically active men

Exclusion Criteria:

* Diabetes, hypertension, obesity subjects, drug use

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the changes of oxidative stress, microcirculation parameters, inflammation biomarkers and plasma adipokines in vitis vinifera extract supplemented and placebo subject before and after high intense training | This study will last 24 months (2013-2015)

SECONDARY OUTCOMES:
Differences between body composition and microcirculation parameters in vitis vinifera extract supplemented and placebo subject before and after high intense training | This study will last 24 months (2013-2015)
Differences between oxidative stress biomarkers in vitis vinifera extract supplemented and placebo subject before and after high intense training | This study will last 24 months (2013-2015)
Differences between inflammation biomarkers in vitis vinifera extract supplemented and placebo subject before and after high intense training | This study will last 24 months (2013-2015)
Differences between adipokines in vitis vinifera extract supplemented and placebo subject before and after high intense training | This study will last 24 months (2013-2015)

CONTACTS AND LOCATIONS:
Overall Officials: J C Koury, PhD, Principal Investigator — Instituto de Nutrição Universidade do Estado do Rio de Janeiro - Brazil
Locations (1):
- Universidade do Estado do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil